CLINICAL TRIAL: NCT05551312
Title: Mobile Virtual Simulation Training in Essential Newborn Care for Healthcare Workers in Low and Middle Income Countries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Lagos, Nigeria (Other); eHealth4everyone (Unknown)
Responsible Party: Principal Investigator, Rachel Umoren, Associate Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00013179; 1R21HD107984 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-09-22 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Resuscitation
Keywords: neonatal; resuscitation; education; virtual; simulation; mobile; phone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Virtual Essential Newborn Care (vENC) Training
  Interventions: Other: Virtual Essential Newborn Care (vENC) training
- Control (No Intervention): Standard of Care

INTERVENTIONS:
Other: Virtual Essential Newborn Care (vENC) training — Essential Newborn Care Mobile Virtual Reality Simulation
  Arms: Intervention

SUMMARY:
Intrapartum asphyxia and prematurity are the leading causes of neonatal mortality in low and middle income countries. Neonatal resuscitation training reduces asphyxia-related newborn mortality and morbidity, but in the absence of continuing low-dose, high frequency practice, these initial gains rapidly decay. The investigators propose to develop and evaluate innovative mobile virtual simulations for refresher training on neonatal resuscitation and essential newborn care to support the retention of knowledge and skills among health care workers in low and middle income countries.

DETAILED DESCRIPTION:
The main goal of this study is to improve newborn mortality and morbidity by using affordable and accessible mobile virtual simulations to provide quality skills training and maintenance for healthcare workers in Low/Middle income countries (LMIC). The investigators hypothesize that mobile devices will provide a readily accessible, standardized alternative to in-person training to maintain skills. This study has the following Specific Aims:

Specific Aim 1: Co-develop and pilot test the usability and efficacy of mobile virtual simulations on early newborn care skills among healthcare workers who attend deliveries in community and health facility-based settings.

Specific Aim 2: Evaluate the impact of the mobile virtual essential newborn care (vENC) training on neonatal resuscitation and care educational indicators and performance outcomes among healthcare workers who provide newborn care in community and health facility-based settings.

Specific Aim 3: Evaluate the impact of virtual simulation refresher training on the rates of neonatal mortality in primary, secondary and tertiary healthcare facilities in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Must have a direct clinical role related to newborn care
* Is able and willing to attend and complete study-related engagements

Exclusion Criteria:

* Healthcare workers who have received essential newborn care course (ENCC) training within the past 12 months at time of recruitment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with correct performance on essential newborn care objective structured clinical exam (OSCE) items at 6 months | at 6 months after in-person training
Early neonatal mortality | within 7 days of birth
  Defined as neonatal mortality within 7 days of birth

SECONDARY OUTCOMES:
Number of participants with correct performance on essential newborn care objective structured clinical exam (OSCE) items by 12 months | at 12 months after in-person training
Number of non-breathing newborns receiving bag and mask ventilation | at delivery
Number of newborns receiving recommended essential newborn care practices | within 7 days of birth
  WHO essential newborn care practices include skin to skin immediately after birth, cord care, early breastfeeding and vitamin K administration
Intrapartum-related mortality | on day 1
  Defined as intrapartum stillbirth (no breathing 10 minutes after delivery)
Early neonatal mortality among babies requiring resuscitation | within 7 days of birth
  Defined as neonatal mortality within 7 days of birth among babies requiring resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Umoren, Principal Investigator — University of Washington
Locations (1):
- University of Lagos, Lagos, Nigeria